CLINICAL TRIAL: NCT03926039
Title: The Effectiveness of Sharing Decision-making Program Interventions in the Early Stage of HCC to Reduce Treatment Decisions Conflicts and Improving Decision-making Satisfaction
Brief Title: Sharing Decision-making Program for HCC Patients Treatment Decisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Lotung Poh-Ai Hospital (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, RN PhD professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CMUH108-REC3-002
Record Dates: First submitted 2019-04-16; First posted 2019-04-24 (Actual); Results first posted 2021-04-15 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Cancer
Keywords: Hepatocarcinoma; sharing decision-making; Health Literacy; decisional conflicts
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Blocked Randomization is a common disease in patients with liver cancer. In order to avoid excessive concentration of the patient control group and the experimental group, the mining blocks are randomly assigned.
Who Masked: Participant
Masking Description: Blocked Randomization is a common disease in patients with liver cancer. In order to avoid excessive concentration of the patient control group and the experimental group, the mining blocks are randomly assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sharing decision-making program interventions (Experimental): Description of conventional traditional treatment options and add sharing decision-making program The intervention measures in this study "sharing decision-making plan" mainly includes sharing the decision-making talks and the decision-making assistance tools used in the process.
  Interventions: Behavioral: sharing decision-making program
- Description of traditional treatment options (No Intervention): Description of conventional traditional treatment options

INTERVENTIONS:
Behavioral: sharing decision-making program — Sharing decision-making talks and decision-making assistance tools used in the process
  Arms: sharing decision-making program interventions

SUMMARY:
Aim: Explore the effectiveness of sharing decision-making program interventions in the early stage of HCC to reduce treatment decisions conflicts and improving decision-making satisfaction.

Design: An experimental design will be used in the study. The 102 primary liver cancer patients, who were diagnosed with Barcelona stage(BCLC stage) 0-A, will be recruited and randomized to the control or intervention group. The intervention measures in this study "sharing decision-making plan" mainly includes sharing the decision-making talks and the decision-making assistance tools used in the process.

DETAILED DESCRIPTION:
The effectiveness of sharing decision-making program interventions in the early stage of HCC to reduce treatment decisions conflicts and improving decision-making satisfactionHepatocarcinoma (HCC) is a high incidence and high mortality disease. Hepatocarcinoma is also a very common disease in Taiwan. Treatment options are limited to those patients with advanced Hepatocarcinoma. However, there are many options for patients with compensated cirrhosis, and small liver tumors are potentially resectable. When patients understood the detailed assessment of the disease both doctors and patients can set the best treatment goals. Sharing decision-making is a patient-centered collaborative processes that enable individuals and their healthcare providers to make decisions together, but patient engagement appears to be less optimistic and there is a lack of evidence that the link between sharing decision-making measures and patient behavior and health outcomes. When decisions are made under social stress or time constraints, people may make less than optimal decisions when they lack sufficient information or skills. Since then the treatment does not match the expected results, often result in decision regrets or arguments with the medical team, and even evolved into medical lawsuits. Therefore, the purpose of this study is to explore the effectiveness of sharing decision-making program interventions in the early stage of HCC to reduce treatment decisions conflicts and improving decision-making satisfaction. In this study, investigators took the experimental design to assess the cases of early hepatocellular carcinoma in hepato- gastroenterology, surgery and oncology clinical in a teaching hospital in the eastern part of Taiwan.

The intervention measures in this study "sharing decision-making plan" mainly includes sharing the decision-making talks and the decision-making assistance tools used in the process. According to Elwyn et.al. (2012), the decision-sharing model was proposed to intervene in the treatment decision-making of early liver cancer patients, including Choice talk, Option talk, Decision talk, and decision-making. Decision support for the process, where the investigator meets with the patient and its important others in the interdisciplinary discussion room or ward meeting room.

Second, decision assistance tools. Decision assistance tools provide information about options and outcomes, and clarify personal values to help people participate in decision making. The aim is to supplement, rather than replace, medical staff counseling (Collins et al., 2009), and the quality of decision aids is very important. Satisfaction with the use of tools is associated with increased patient satisfaction and reduced decision-making. Patients can benefit from computerized decision-making tools without the need to increase physician involvement.

The research tools include basic population data, clinical stage of disease, self-efficacy scale of hepatocellular carcinoma, Decision Decision Confidence Scale (DCS), decision self-efficacy scale , Decision Satisfaction Scale and Chinese Simplified-form Mandarin Health Literacy Scale.

The obtained data were collected and analyzed by SPSS20.0 for Window software. The main statistical methods include descriptive statistics, T-test, analysis of variance, Pearson Product Moment correlation coefficient and Generalized Estimating Equations (GEEs) ).

ELIGIBILITY:
Inclusion Criteria:

1. Primary liver cancer patients (ICD 10 is C22.0) and Barcelona stage (BCLC stage) 0-A.
2. At least 20 years of age.
3. No mental illness.
4. Patients who can communicate in Mandarin or Taiwanese.

Exclusion Criteria:

1. Don't know himself condition.
2. Unconscious patients.
3. Patients with liver cancer resection or partial liver resection were performed within 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsae Jyy Wang, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Lo-Hsu medical foundation Lotung Poh-Ai hospital, Yilan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Degner LF, Kristjanson LJ, Bowman D, Sloan JA, Carriere KC, O'Neil J, Bilodeau B, Watson P, Mueller B. Information needs and decisional preferences in women with breast cancer. JAMA. 1997 May 14;277(18):1485-92. PMID 9145723
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Background] Bruix J, Reig M, Sherman M. Evidence-Based Diagnosis, Staging, and Treatment of Patients With Hepatocellular Carcinoma. Gastroenterology. 2016 Apr;150(4):835-53. doi: 10.1053/j.gastro.2015.12.041. Epub 2016 Jan 12. PMID 26795574
- [Background] Katie Lee SY, Knobf MT. Primary Breast Cancer Decision-making Among Chinese American Women: Satisfaction, Regret. Nurs Res. 2015 Sep-Oct;64(5):391-401. doi: 10.1097/NNR.0000000000000116. PMID 26325281
- [Derived] Liao YL, Wang TJ, Su CW, Liang SY, Liu CY, Fan JY. Efficacy of a Decision Support Intervention on Decisional Conflict Related to Hepatocellular Cancer Treatment: A Randomized Controlled Trial. Clin Nurs Res. 2023 Jan;32(1):233-243. doi: 10.1177/10547738221121447. Epub 2022 Sep 8. PMID 36082423

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After screening for inclusion and exclusion criteria, cases eligible for admission were recruited, and the researcher explained the research purpose and steps to the research subjects in the clinic room and completed the consent form after the patient agreed to participate in the study. Randomly assigned to control or experimental groups
Period: Overall Study
Arm/Group | Sharing Decision-making Program Interventions | Description of Traditional Treatment Options
Started | 35 | 35
Completed | 35 | 34
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 72 people are eligible for recruitment criteria. One person was transferred to the medical center hospital and refused to participate. Another person did not know the condition and therefore excluded. A total of 70 participants randomly allocated to the intervention group and control group. There is one participant who was a dropout due to go to a medical center for surgery. The effective sample was 69.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sharing Decision-making Program Interventions | Description of Traditional Treatment Options | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (11.3) | 67.1 (13.5) | 65.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 24 | 22 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 35 | 34 | 69
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 35 | 34 | 69
BCLC stage [Count of Participants; unit: Participants] — Barcelona clinic liver cancer (BCLC) staging uses a set of criteria to guide the management of patients with hepatocellular carcinoma (HCC).stage 0 (very early stage);stage A (early stage);stage B (intermediate stage)
  Participants
    BCLC stage 0 (very early stage) | 12 | 14 | 26
    BCLC stage A (early stage) | 19 | 14 | 33
    BCLC stage B (intermediate stage) | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Decisional Conflict Scale
Description: 5 questions for a total of 16 questions, respectively, to assess the uncertainty of the subscale (10-12 questions) the subscale total score range 0-300 points , informed subscales (1-3 questions) the subscale total score range 0-300 points, values subscales (4-6 questions) the subscale total score range 0-300 points, support subscales ( 7-9 questions) the subscale total score range 0-300 points, effective decision-making scale (13-16 questions) the subscale total score range 0-300 points, Each question is scored on a Likert scale of 0-4 points (very strongly agreed to very disagree), then multiplied by 25 so that each question may score 0-100 points. A score of 0 is a good decision, and a score of 100 is the worst decision. the total score was 0 to 1600 points.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sharing Decision-making Program Interventions | Description of Traditional Treatment Options
Number analyzed (Participants) | 35 | 34
score on a scale | 6.9 (9.7) | 11 (14.3)
Statistical Analysis 1: Comparison: Sharing Decision-making Program Interventions vs Description of Traditional Treatment Options; Both group of average difference (95% CI) in intervention group and control group; Test type: Equivalence — Equivalence Analysis; p = 0.05, ANOVA

2. Secondary Outcome: Satisfaction With Decision Instrument
Description: The content consists of 6 items, with a score of 1-5 points (very strongly disagreed and very agreeable) for each question. The score may be 6-30 points. The higher the score, the higher the satisfaction with the decision. A score of 6 indicates that the extreme dissatisfaction of 30 points indicates extreme satisfaction.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sharing Decision-making Program Interventions | Description of Traditional Treatment Options
Number analyzed (Participants) | 35 | 34
score on a scale | 26.2 (2.2) | 27.1 (3.3)

3. Secondary Outcome: Decision Self-efficacy Scale
Description: The scale included 11 questions, and participants were asked to think about how confident they were in making informed choices in 11 situations. The scoring for each situation is scored on a Likert scale with 0-4 points (very agrees to very disagree) for each question, then multiplied by 25 so that each question may score 0-100 points. The higher the score, the more confident participant are. Each question 0 points is not confident, 100 points is very confident. total score range is 0- 1100 points
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sharing Decision-making Program Interventions | Description of Traditional Treatment Options
Number analyzed (Participants) | 35 | 34
score on a scale | 73.3 (11.4) | 72.1 (15.6)

4. Secondary Outcome: Liver Cancer Treatment Options Related Knowledge Scale
Description: A total of 20 questions total score of 100 points, the higher the knowledge, the better.Total scale range was 5-100 points.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sharing Decision-making Program Interventions | Description of Traditional Treatment Options
Number analyzed (Participants) | 35 | 34
score on a scale | 84.6 (13.3) | 75.6 (6.8)

5. Other Pre Specified Outcome: Control Preference Scale
Description: The scale is patients make treatment decisions in life-threatening conditions. For the first time, ask patients about their preferred clinical decision-making role. Then, ask a second time for the style they experienced. The instrument doesn't have any score on a scale. Each question was counted independently, the maximum is the number of participants in each group. the minimum is zero.
Time Frame: 1 week
Measure: Number; unit: Count of Participants
Arm/Group | Sharing Decision-making Program Interventions | Description of Traditional Treatment Options
Number analyzed (Participants) | 34 | 34
Count of Participants
  I hope that I have seriously considered the opinions of the doctor and let me make my own decisions | 13 | 11
  I hope that the doctor and I together making decisions | 9 | 11
  I hope that my doctor will make the final decision on the treatment | 6 | 5
  I prefer my doctor to make all related treatment decisions | 7 | 7

6. Other Pre Specified Outcome: Decision Regret Scale
Description: The DRS was used to evaluate the feeling of regret after making a decision. There are 5 questions on the scale. The scoring of each situation is based on a Likert scale of 1-5 points (from strongly agree to strongly disagree) for each question. The score is subtracted by 1 and then multiplied by 25, so that each question may be scored 0-100 Minute. The final score is added and averaged. The score range is 0-100 points. The higher the score, the more regretful it is, the 0 point means no regret and 100 points means very regret.
Time Frame: around 3 month after discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sharing Decision-making Program Interventions | Description of Traditional Treatment Options
Number analyzed (Participants) | 35 | 34
score on a scale | 20 (12.2) | 22.4 (13.5)

ADVERSE EVENTS:
Time Frame: around 3 month
Arm/Group | Sharing Decision-making Program Interventions | Description of Traditional Treatment Options
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

LIMITATIONS AND CAVEATS:
The participants' average age of onset was 65 years old, and the education level was below the elementary school. Some cases need to be read verbatim and assisted in checking. , Maybe slightly different from the self-reading, but the researchers still try to be neutral and consistent when reading the questionnaire, so as not to affect the participants' answers

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT03926039/Prot_SAP_000.pdf